CLINICAL TRIAL: NCT00907959
Title: A Phase 2 Clinical Trial Assessing Safety and Efficacy of BZL101 for Metastatic Breast Cancer
Brief Title: A Clinical Trial Assessing Safety and Efficacy of BZL101 for Metastatic Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bionovo (Industry)
Responsible Party: Mary Tagliaferri, Chief Medical Officer, Bionovo
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BZL-101-003
Record Dates: First submitted 2009-05-22; First posted 2009-05-25 (Estimated); Last update posted 2012-02-08 (Estimated); Status verified 2012-02

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Scutellaria barbata extract

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: BZL101 — Oral BZL101 20 grams/day (10 grams BID).

SUMMARY:
The investigators' proposed phase 2 clinical trial will be an open-label, non-randomized study among 80 women with metastatic breast cancer. The study treatment period will be up to twelve months and enrollment will be open at 10-15 clinical sites in the United States. In this Phase 2 trial, 40 participants with hormone receptor positive tumors and 40 with hormone receptor negative tumors will be enrolled and treated with BZL101 20 grams/day (10 grams BID). Hormone receptor positive will be defined as estrogen receptor (ER)+ and progesterone receptor (PR)+, ER+ and PR-, or ER- and PR+. Hormone receptor negative will be defined as ER- and PR-.

ELIGIBILITY:
Inclusion Criteria:

1. Women 18 years or older.
2. Histologically confirmed diagnosis of breast cancer based on pathology report of primary, regional or metastatic breast cancer.
3. Clinical evidence of metastatic (stage IV) involvement other than bone only metastasis based on the investigator's clinical and/or radiographic findings.
4. Availability of estrogen receptor and progesterone receptor status measured on biopsy tissue. (Status on the most recent biopsy where ER/PR status was documented will be used to determine hormone receptor status for stratification).
5. At least one measurable disease site defined by RECIST criteria, with measurement made within 30 days of beginning study therapy. (Non-measurable disease includes bone lesions, leptomeningeal disease, ascites, pleural/pericardial effusion, inflammatory breast disease, lymphangitis cutis/pulmonis, abdominal masses that are not confirmed and followed by imaging techniques, and cystic lesions. For lesions in a previously irradiated field, the radiated lesion cannot be assessed as a measurable lesion unless growth of that lesion has been documented after radiation).
6. No more than 2 prior cytotoxic regimens administered for metastatic breast cancer. (Participants may have received any number of exogenous hormone therapies for Stage IV disease and/or adjuvant therapy).
7. Life expectancy of >12 weeks.
8. Eastern Cooperative Oncology Group performance status <2.
9. Women of child bearing potential must agree to use two adequate methods of contraception or abstain from sexual intercourse during study treatment. Acceptable methods of contraception are as follows:

   1. Intrauterine device (IUD)
   2. Hormonal birth control
   3. Tubal ligation
   4. Partner's vasectomy
   5. Latex condom
   6. Diaphragm
   7. Cervical cap
10. Adequate organ and marrow function measured within 14 days of study treatment as defined below:

Absolute neutrophil count >1,500 cells/mm3 Platelets >100,000 cells/mm3 Hemoglobin >10 g/dL Total bilirubin <1.5 mg/dL AST(SGOT)/ALT(SGPT) <2.5 X institutional upper limit of normal or <5 X normal with documented liver metastasis Alkaline Phosphatase <3 X institutional upper limit of normal or <5 X normal with documented liver or bone metastasis Serum creatinine <1.5 mg/dL or Creatinine clearance >60 mL/min/1.73 m2 for participants with serum creatinine levels above institutional normal.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2012-01; Primary Completion 2015-01 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
The primary outcomes of the Phase 2 trial will be safety and toxicity as measured by NCI Common Terminology Criteria for Adverse Events (CTCAE), Version 4.0 and tumor response rate defined by new RECIST criteria 1.1. | Monthly

CONTACTS AND LOCATIONS:
Locations (1):
- M.D. Anderson Cancer Center, Houston, Texas, United States